CLINICAL TRIAL: NCT03136445
Title: A Double-blind, Randomised Controlled Trial Evaluating the Safety and Efficacy of Antifibrinolytics (Tranexamic Acid) in Patients With Haematological Malignancies With Severe Thrombocytopenia
Brief Title: TRial to EvaluAte Tranexamic Acid Therapy in Thrombocytopenia
Acronym: TREATT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NHS Blood and Transplant (Other Government)
Collaborators: National Health and Medical Research Council, Australia (Other); Monash University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 12-01-CSU; 2014-001513-35 (EudraCT Number); ISRCTN73545489 (Registry Identifier: ISRCTN Registry)
Record Dates: First submitted 2017-02-21; First posted 2017-05-02 (Actual); Results first posted 2025-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-09

CONDITIONS: Hematologic Neoplasms; Hemorrhage; Hematopoietic Stem Cell Transplantation
Keywords: Tranexamic acid; Platelet transfusion
MeSH Terms: conditions — Hematologic Neoplasms; Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Arm (Experimental): Tranexamic acid (TXA). Dose schedule TXA 1g every eight hours IV or 1.5g every eight hours PO.
  Interventions: Drug: Tranexamic acid (TXA).
- Control Arm (Placebo Comparator): Placebo (saline) if administration is IV. Placebo tablet matched for appearance to TXA if oral.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic acid (TXA). — IV or oral preparation. IV tranexamic acid or Oral tablet of tranexamic acid.
  Other Names: Cyklokapron®; trans-4-(aminomethyl)cyclohexanecarboxylic acid; Lysteda
  Arms: Intervention Arm
Drug: Placebo — IV (saline) or oral placebo tablets
  Other Names: Placebo for tranexamic acid
  Arms: Control Arm

SUMMARY:
The purpose of this study is to test whether giving tranexamic acid to patients receiving treatment for blood cancers reduces the risk of bleeding or death, and the need for platelet transfusions. Patients will be randomised to receive tranexamic acid (given intravenously through a drip, or orally) or a placebo.

DETAILED DESCRIPTION:
Patients with cancers of the blood often develop low blood cell counts either as a consequence of the disease or the treatment by chemotherapy or stem cell transplantation. Platelet transfusions are commonly given to raise any low platelet count and reduce the risk of clinical bleeding (prophylaxis) or stop active bleeding (therapy). But recent studies have indicated that many patients continue to experience bleeding, despite the use of platelet transfusions. Tranexamic acid is a type of drug that is called an antifibrinolytic. These drugs act to reduce the breakdown of clots formed in response to bleeding. These drugs have been used widely in both elective and emergency surgery and have been shown to decrease blood loss and the use of red cell transfusions. The purpose of this study is to test whether giving tranexamic acid to patients receiving treatment for blood cancers reduces the risk of bleeding or death, and the need for platelet transfusions. Patients will be randomised to receive tranexamic acid (given intravenously through a drip, or orally) or a placebo. The investigators will measure the rates of bleeding daily using a short structured assessment of bleeding and will record the number of transfusions given to patients.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible for this trial if:

1. Aged ≥18 years of age
2. Confirmed diagnosis of a haematological malignancy
3. Undergoing chemotherapy, or chemotherapy is planned, or haematopoietic stem cell transplantation
4. Anticipated to have a hypoproliferative thrombocytopenia resulting in a platelet count of ≤10x10⁹/L for ≥ 5 days
5. Able to comply with treatment and monitoring

Exclusion Criteria:

A patient will not be eligible for this trial if he/she fulfils one or more of the following criteria:

1. Patients with a past history or current diagnosis of arterial or venous thromboembolic disease including myocardial infarction, peripheral vascular disease and retinal arterial or venous thrombosis.
2. Diagnosis of acute promyelocytic leukaemia (APML) and undergoing induction chemotherapy
3. Patients with a diagnosis/previous history of veno-occlusive disease (also called sinusoidal obstruction syndrome)
4. Patients with known inherited or acquired prothrombotic disorders e.g.

   1. Lupus anticoagulant
   2. Positive antiphospholipids
5. Patients receiving any pro-coagulant agents (e.g. DDAVP, recombinant Factor VIIa or Prothrombin Complex Concentrates (PCC) within 48 hours of enrolment, or with known hypercoagulable state
6. Patients receiving L-asparaginase as part of their current cycle of treatment
7. History of immune thrombocytopenia (ITP), thrombotic thrombocytopenic purpura (TTP) or haemolytic uraemic syndrome (HUS)
8. Patients with overt disseminated intravascular coagulation (DIC) (See Appendix 3 in the protocol for definition)
9. Patients requiring a platelet transfusion threshold >10x10/⁹L at time of randomisation. (This refers to patients who require their platelet count to be maintained at a certain specified level on an ongoing basis, and excludes a transient rise in the threshold due to sepsis.)
10. Patients with a known inherited or acquired bleeding disorder e.g.

    1. Acquired storage pool deficiency
    2. Paraproteinaemia with platelet inhibition
11. Patients receiving anticoagulant therapy or anti-platelet therapy
12. Patients with visible haematuria at time of randomisation
13. Patients with anuria (defined as urine output < 10 mls/hr over 24 hours).
14. Patients with severe renal impairment (eGFR ≤30 ml/min/1.73m²)
15. Patients with a previous history of epilepsy, convulsions, fits or seizures
16. Patients who are pregnant or breast-feeding
17. Allergic to tranexamic acid.
18. Patients enrolled in other trials involving platelet transfusions, anti-fibrinolytics, platelet growth factors or other pro-coagulant agents.
19. Patients previously randomised into this trial at any stage of their treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lise J Estcourt, MBBChir MSc DPhil MRCP FRCPath, Principal Investigator — NHS Blood and Transplant; Zoe K McQuilten, MBBS PhD, Principal Investigator — Monash University; Simon J Stanworth, DPhil FRCP FRCPath, Principal Investigator — NHS Blood and Transplant; Erica M Wood, MB BS, FRACP, FRCPA, Principal Investigator — Monash University
Locations (27):
- Australia (11):
  - Royal Adelaide Hospital, Adelaide
  - Royal Brisbane, Brisbane
  - Canberra Hospital, Canberra
  - Andrew Love Cancer Centre, Geelong
  - Alfred Hospital, Melbourne
  - Monash Health, Melbourne
  - St Vincent's Hospital, Melbourne
  - Victorian Comprehensive Cancer Centre, Melbourne
  - Royal North Shore Hospital, St Leonards
  - St Vincent's Hospital, Sydney
  - Westmead Hospital, Westmead
- United Kingdom (16):
  - Royal United Hospital, Bath
  - Belfast City Hospital, Belfast
  - Heartlands Hospital, Birmingham
  - Queen Elizabeth Hospital, Birmingham
  - Bristol Haematology and Oncology Centre, Bristol
  - University Hospital Coventry, Coventry
  - Royal Devon and Exeter Hospital, Exeter
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St James's Hospital, Leeds
  - Lincoln County Hospital, Lincoln
  - King's College Hospital, London
  - University College London Hospitals, London
  - Freeman Hospital, Newcastle
  - Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth
  - Salisbury District Hospital, Salisbury

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analysed during the current study will be available upon request from the NHSBT Clinical Trials Unit after de-identification (text, tables, figures and appendices) 9 months after publication and ending 5 years following article publication.
Supporting Information: Study Protocol
Time Frame: 9 months after publication and ending 5 years following article publication.
Access Criteria: Data will be shared with investigators whose use of the data has been assessed and approved by an NHSBT review committee as a methodologically sound proposal.

REFERENCES:
- [Result] TREATT Trial Investigators. Tranexamic acid versus placebo to prevent bleeding in patients with haematological malignancies and severe thrombocytopenia (TREATT): a randomised, double-blind, parallel, phase 3 superiority trial. Lancet Haematol. 2025 Jan;12(1):e14-e22. doi: 10.1016/S2352-3026(24)00317-X. Epub 2024 Dec 3. PMID 39642900
- [Derived] Estcourt LJ, McQuilten Z, Powter G, Dyer C, Curnow E, Wood EM, Stanworth SJ; TREATT Trial Collaboration (provisional). The TREATT Trial (TRial to EvaluAte Tranexamic acid therapy in Thrombocytopenia): safety and efficacy of tranexamic acid in patients with haematological malignancies with severe thrombocytopenia: study protocol for a double-blind randomised controlled trial. Trials. 2019 Oct 15;20(1):592. doi: 10.1186/s13063-019-3663-2. PMID 31615553
- See also: Published paper- Tranexamic acid versus placebo to prevent bleeding in patients with haematological malignancies and severe thrombocytopenia (TREATT): a randomised, double-blind, parallel, phase 3 superiority trial — https://doi.org/10.1016/S2352-3026(24)00317-X
- Available data/document: Study Protocol: PMC6792262 — https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-019-3663-2 — The protocol was published in The Trials Journal, The TREATT Trial (TRial to EvaluAte Tranexamic acid therapy in Thrombocytopenia): safety and efficacy of tranexamic acid in patients with haematological malignancies with severe thrombocytopenia: study protocol for a double-blind randomised controlled trial. Trials Free Article - Estcourt LJ, McQuilten Z, Powter G, Dyer C, Curnow E, Wood EM, Stanworth SJ, TREATT Trial Collaboration (provisional). To request a protocol please contact the Trial Manager Gillian Powter gillian.powter@nhsbt.nhs.uk

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm | Control Arm
Started | 310 | 306
Completed | 300 | 297
Not Completed | 10 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 310 | 306 | 616
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 1 participant missing this information
  years
    number analyzed (Participants) | 309 | 306 | 615
    (all) | 55.8 (12.3) | 55.3 (12.1) | 55.6 (12.2)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: 1 participant missing this information
  Participants
    number analyzed (Participants) | 309 | 306 | 615
    Male | 194 | 186 | 380
    Female | 115 | 120 | 235
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 272 | 266 | 538
  Asian | 7 | 14 | 21
  Black African | 1 | 1 | 2
  Black Caribbean | 2 | 1 | 3
  Arab / Other Middle East ancestry | 1 | 3 | 4
  Aboriginal | 2 | 1 | 3
  Other | 4 | 5 | 9
  Unknown / Not Stated | 17 | 13 | 30
  (Mixed ethnic group:) White / Black Caribbean | 2 | 0 | 2
  (Mixed ethnic group:) White / Other | 1 | 1 | 2
  (Mixed ethnic group:) Other mixed ethnic group | 1 | 1 | 2
Height [Mean (Standard Deviation); unit: cm] — Population: 6 participants missing this information
  cm
    number analyzed (Participants) | 305 | 305 | 610
    (all) | 172.4 (10.1) | 171.7 (9.7) | 172.1 (9.9)
Weight [Mean (Standard Deviation); unit: kg] — Population: 4 participants missing this information
  kg
    number analyzed (Participants) | 307 | 305 | 612
    (all) | 81.1 (16.6) | 80.5 (17.6) | 80.8 (17.1)
Diagnosis [Count of Participants; unit: Participants] — Population: 1 participant missing this information
  Participants
    number analyzed (Participants) | 309 | 306 | 615
    AML | 135 | 129 | 264
    ALL | 9 | 11 | 20
    APL | 0 | 2 | 2
    CML | 5 | 7 | 12
    CLL | 3 | 4 | 7
    Hodgkin's Lymphoma | 17 | 12 | 29
    Non-Hodgkin Lymphoma | 70 | 62 | 132
    Myeloma | 35 | 36 | 71
    MDS | 18 | 22 | 40
    Other | 17 | 21 | 38
Treatment plan [Count of Participants; unit: Participants] — Population: 1 participant missing this information
  Participants
    number analyzed (Participants) | 309 | 306 | 615
    Induction chemotherapy | 70 | 72 | 142
    Consolidation chemotherapy | 49 | 46 | 95
    Autograft | 111 | 105 | 216
    Allograft | 77 | 79 | 156
    Other | 2 | 4 | 6
Platelet count at consent [Mean (Standard Deviation); unit: 10^9 cells/L] — Population: 4 participants missing this information
  10^9 cells/L
    number analyzed (Participants) | 309 | 303 | 612
    (all) | 116.2 (103.3) | 113.1 (94.9) | 114.7 (99.1)
Platelet count at randomisation [Mean (Standard Deviation); unit: 10^9 cells/L] — Population: 3 participants missing this information
  10^9 cells/L
    number analyzed (Participants) | 309 | 304 | 613
    (all) | 31.7 (18.1) | 29.2 (13.3) | 30.4 (15.9)
Haemoglobin at consent [Mean (Standard Deviation); unit: G/L] — Population: 5 participants missing this information
  G/L
    number analyzed (Participants) | 308 | 303 | 611
    (all) | 100.2 (18.1) | 98.5 (18) | 99.4 (18)
Haemoglobin at randomisation [Mean (Standard Deviation); unit: G/L] — Population: 3 participants missing this information
  G/L
    number analyzed (Participants) | 309 | 304 | 613
    (all) | 94.3 (16) | 91.2 (15.8) | 92.8 (15.9)
FACT-G subscale score at randomisation [Mean (Standard Deviation); unit: scores on a scale] — Functional Assessment of Cancer Therapy General (FACT-G)
  Description: General quality of life instrument intended for use with a variety of chronic illness conditions.
  Number of items: 27 (7 for each category, excluding emotional which is 6)
  Name of categories/domains: Physical, social/family, emotional, and functional well-being.
  Scoring: Subscale scores added to obtain category scores.
  Interpretation: A higher total score demonstrates a better quality of life. (Physical, social/family, functional well-being score range: 0-28, Emotional score range: 0-24) Population: Some participants are missing data for these QOL questionnaires
  scores on a scale
    Physical well-being: number analyzed (Participants) | 272 | 278 | 550
    Physical well-being | 16.4 (7.1) | 17.1 (6.7) | 16.7 (6.9)
    Social/family well-being: number analyzed (Participants) | 272 | 278 | 550
    Social/family well-being | 23.8 (4.7) | 23.7 (4.5) | 23.7 (4.6)
    Emotional well-being: number analyzed (Participants) | 271 | 275 | 546
    Emotional well-being | 18.3 (4.1) | 18.5 (4.3) | 18.4 (4.2)
    Functional well-being: number analyzed (Participants) | 270 | 272 | 542
    Functional well-being | 14.3 (6.2) | 14.3 (6.8) | 14.3 (6.5)
FACT-G total score at randomisation [Mean (Standard Deviation); unit: scores on a scale] — Functional Assessment of Cancer Therapy General (FACT-G)
  Description: General quality of life instrument intended for use with a variety of chronic illness conditions.
  Scoring: Category scores added to obtain total score.
  Interpretation: A higher total score demonstrates a better quality of life. (FACT-G total score range: 0-108) Population: 76 participants missing this information
  scores on a scale
    number analyzed (Participants) | 268 | 272 | 540
    (all) | 72.6 (14.5) | 73.6 (16.6) | 73.1 (15.6)
FACT-Th total score at randomisation [Mean (Standard Deviation); unit: scores on a scale] — Functional Assessment of Cancer Therapy - Thrombocytopenia (18-item version) (FACT-Th18)
  Objective: To measure the self-reported quality of life (QoL) concerns of patients with thrombocytopenia
  Interpretation: A higher total score demonstrates a better quality of life (FACT-Th total score range: 0-180) Population: 79 participants missing this information
  scores on a scale
    number analyzed (Participants) | 266 | 271 | 537
    (all) | 125.7 (22) | 127.6 (24.5) | 126.7 (23.3)
Medical history [Count of Participants; unit: Participants] — Population: Some participants are missing data for medical history
  Participants
    Diabetes requiring treatment: number analyzed (Participants) | 309 | 306 | 615
    Diabetes requiring treatment | 21 | 20 | 41
    Hypertension requiring treatment: number analyzed (Participants) | 309 | 306 | 615
    Hypertension requiring treatment | 42 | 40 | 82
    Renal impairment requiring treatment: number analyzed (Participants) | 309 | 306 | 615
    Renal impairment requiring treatment | 6 | 5 | 11
    Confirmed invasive fungal infection: number analyzed (Participants) | 309 | 306 | 615
    Confirmed invasive fungal infection | 10 | 3 | 13
    Other malignancy: number analyzed (Participants) | 309 | 306 | 615
    Other malignancy | 10 | 8 | 18
    HLA antibodies: number analyzed (Participants) | 307 | 306 | 613
    HLA antibodies | 1 | 6 | 7

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients Who Die or Have Bleeding of WHO Grade 2 or Above by WHO Criteria During the First 30 Days From the First Dose of Trial Treatment, or Planned First Dose for Those Participants Who do Not Receive Treatment.
Description: The proportion of patients who die or have bleeding of WHO grade 2 or above by WHO criteria during the first 30 days from the first dose of trial treatment, or planned first dose for those participants who do not receive treatment.
  A time-to-event analysis will be used to determine this proportion to ensure that all patients are included in the primary outcome analysis, not just those who are followed up for the full 30 days. Any patients lost to follow-up will be included in the analysis and censored at the time that they were lost.
Time Frame: The first 30 days from first dose of trial treatment
Population: Participants with primary outcome data reported
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 298 | 295
percentage of participants | 31.7 [26.6 to 37.4] | 34.2 [29.0 to 40.0]

2. Secondary Outcome: Mean (SD) Percentage of Days With WHO Grade 2 Bleeding or Above, Per Participant.
Description: Number of days where WHO grade 2 or above bleeding has been recorded bleeding using WHO bleeding criteria.
Time Frame: The first 30 days from first dose of trial treatment .
Population: Participants with primary outcome data reported
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 298 | 295
percentage of days | 3.1 (9.5) | 3.2 (7.8)

3. Secondary Outcome: Time to First Episode of Bleeding of WHO Grade 2 or Greater up to Study Day 30.
Description: Bleeding assessed using WHO bleeding criteria. Time to first episode of bleeding of WHO grade 2 or above was estimated using a cumulative incidence function, with death as a competing risk. The lower quartile for the time is reported as the median was not estimable.
Time Frame: The first 30 days from first dose of trial treatment.
Population: Participants with primary outcome data reported
Measure: Median (Inter-Quartile Range); unit: Lower quartile for number of days
Units Other Than Participants: Days
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 298 | 295
Number analyzed (Days) | 30 | 30
Lower quartile for number of days | NA [10.5 to NA] — Median is not estimable due to insufficient number of events | NA [8.5 to NA] — Median is not estimable due to insufficient number of events

4. Secondary Outcome: Highest Grade of Bleeding a Patient Experiences up to Study Day 30.
Description: Measured using WHO bleeding criteria (The higher the grade, the most severe the bleed).
  Grade 0: no bleeding Grade 1: petechial bleeding Grade 2: mild blood loss (clinically significant) Grade 3: gross blood loss, requires transfusion(severe) Grade 4: debilitating blood loss, retinal or cerebral associated with fatality
Time Frame: The first 30 days from first dose of trial treatment.
Population: Data is only presented for participants who experienced at least one bleed
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 205 | 225
Participants
  Grade 0 | 7 | 6
  Grade unassigned | 0 | 1
  Grade 2 | 85 | 93
  Grade 3 | 0 | 3
  Grade 4 | 2 | 1
  Grade 1 | 111 | 121

5. Secondary Outcome: Number of Platelet Transfusions Per Patient up to Study Day 30.
Description: Measured by number of recorded platelet transfusions per patient.
Time Frame: The first 30 days from first dose of trial treatment.
Population: Participants with primary outcome data reported
Measure: Median (Inter-Quartile Range); unit: platelet units
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 298 | 295
platelet units | 3 [1 to 6] | 3 [1 to 6]

6. Secondary Outcome: Number of Red Cell Transfusions Per Patient up to Study Day 30.
Description: Measured by number of recorded red cell transfusions per patient.
Time Frame: The first 30 days from first dose of trial treatment.
Population: Participants with primary outcome data reported
Measure: Median (Inter-Quartile Range); unit: Red cell units
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 298 | 295
Red cell units | 2 [0 to 4] | 2 [1 to 4]

7. Secondary Outcome: Proportion of Patients Surviving at Least 30 Days Without a Platelet Transfusion.
Description: Measured by calculating number of patients surviving at least 30 days without a platelet transfusion.
Time Frame: The first 30 days from first dose of trial treatment.
Population: Participants with primary outcome data reported
Measure: Number (95% Confidence Interval); unit: proportion
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 298 | 295
proportion | 8.3 [5.4 to 11.9] | 6.4 [3.9 to 9.7]

8. Secondary Outcome: Proportion of Patients Surviving at Least 30 Days Without a Red Cell Transfusion.
Description: Measured by calculating the number of patients surviving at least 30 days without a red cell transfusion.
Time Frame: The first 30 days from first dose of trial treatment.
Population: Participants with primary outcome data reported
Measure: Number (95% Confidence Interval); unit: proportion
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 298 | 295
proportion | 29.4 [24.1 to 34.8] | 20.5 [16.0 to 25.4]

9. Secondary Outcome: Number of Participants With a Thrombotic Event From First Administration of Trial Treatment up to and Including 120 Days After the First Dose of Trial Treatment is Received (N)
Description: Measured by calculating number of patients developing clinically diagnosed thrombotic events within 120 days of Treatment Day 1 i.e the first day that the IMP is administered.
Time Frame: Up to and including 120 days from the first administration of investigational medicinal product (IMP).
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 300 | 297
Participants | 8 | 5

10. Secondary Outcome: Number of Patients Developing Veno-occlusive Disease (VOD; Sinusoidal Obstructive Syndrome, SOS) Within 60 Days of First Administration of Trial Treatment.
Description: Measured by calculating number of patients developing Veno-occlusive Disease (VOD; Sinusoidal obstructive syndrome, SOS) within 60 days of Treatment Day 1 i.e the first day that the IMP is administered.
Time Frame: Up to and including 60 days from the first administration of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 300 | 297
Participants | 3 | 2

11. Secondary Outcome: All-cause Mortality During the First 30 Days and 120 Days After the First Dose of Trial Treatment is Administered.
Description: Measured by calculating number of deaths in first 30 days and 120 days after Treatment Day 1 i.e the first day that the IMP is administered.
Time Frame: Up to and including 120 days from the first administration of IMP.
Population: 4 Participants were missing mortality data and so weren't analysd
Measure: Number (95% Confidence Interval); unit: proportion
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 298 | 295
proportion
  30 days | 2.9 [1.5 to 5.8] | 1.1 [0.4 to 3.3]
  120 days | 8.7 [5.9 to 12.8] | 5.3 [3.2 to 8.8]

12. Secondary Outcome: Death Due to Thrombosis During the First 120 Days After the First Dose of Trial Treatment is Administered.
Description: Measured by calculating number of deaths due to thrombosis during the first 120 days after Treatment Day 1 i.e the first day that the IMP is administered.
Time Frame: Up to and including 120 days from the first administration of IMP.
Measure: Number; unit: percent
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 300 | 297
percent | 0 | 0

13. Secondary Outcome: Death Due to Bleeding During the First 30 Days After the First Dose of Trial Treatment is Administered.
Description: Measured by calculating number of deaths due to bleeding during the first 30 days
Time Frame: Up to and including 30 days from the first administration of IMP.
Measure: Number; unit: percent
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 300 | 297
percent | 0 | 0

14. Secondary Outcome: Number of Serious Adverse Events (SAE) From First Administration of Trial Treatment Until 60 Days After the First Dose of Trial Treatment is Administered.
Description: Measured by calculating the total number of SAE's reported from first administration of IMP.
Time Frame: Up to and including 60 days from the first administration of IMP.
Measure: Number; unit: Serious adverse events
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 300 | 297
Serious adverse events
  Total number of serious adverse events (SAE) up to day 60 | 94 | 103
  Sepsis | 25 | 27
  Organ failure | 4 | 7
  GvHD | 5 | 7
  Transfusion reaction | 2 | 4
  Fever | 24 | 20
  Other SAEs | 34 | 38

15. Other Pre Specified Outcome: Proportion of Days With Thrombocytopenia (≤10x10⁹/L, ≤30x10⁹L, ≤50x10⁹/L).
Description: Measured by number of days that the patient's laboratory results indicate that the patient is thrombocytopenic.
Time Frame: Measured during first 30 days from first dose of IMP.
Population: Days platelet count count was recorded (so risk of thrombocytopenia could be detected)
Measure: Mean (Standard Deviation); unit: Days with thrombocytopenia
Units Other Than Participants: Days a platelet count should be reported
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 298 | 295
Number analyzed (Days a platelet count should be reported) | 5271 | 5326
Days with thrombocytopenia
  Thrombocytopenia (≤10x109/L) | 13.7 (13.9) | 15.3 (15.4)
  Thrombocytopenia (≤30x109/L) | 64.8 (25.9) | 60.2 (24.8)
  Thrombocytopenia (≤50x109/L) | 78.2 (22.3) | 74 (23.1)

16. Other Pre Specified Outcome: Reasons for Platelet Transfusions.
Description: Reasons for platelet transfusions as documented by clinician.
Time Frame: Measured during first 30 days from first dose of IMP.
Population: Participants with at least one platelet transfusion
Measure: Number; unit: Platelet transfusions
Units Other Than Participants: Number of platelet transfusions
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 267 | 275
Number analyzed (Number of platelet transfusions) | 1205 | 1264
Platelet transfusions
  Prophylaxis for platelet count ≤10x109/L | 438 | 456
  Prophylaxis and platelet count >10x109/L | 671 | 705
  Invasive procedure | 27 | 31
  Active bleeding | 59 | 66
  Missing data for reasons for platelet transfusions | 10 | 6

17. Other Pre Specified Outcome: Reasons for Red Cell Transfusions.
Description: Reasons for red cell transfusions as documented by clinician.
Time Frame: Measured during first 30 days from first dose of IMP.
Population: Participants with at least one red cell transfusion
Measure: Number; unit: Red cell transfusions
Units Other Than Participants: Number of red cell transfusions given
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 202 | 230
Number analyzed (Number of red cell transfusions given) | 766 | 845
Red cell transfusions
  Low haemoglobin | 736 | 818
  Active bleeding | 7 | 7
  Other | 17 | 14
  Missing data for reasons for red cell transfusions | 6 | 6

18. Other Pre Specified Outcome: Proportion of Days With Fever
Description: Highest daily temperature ≥ 38.1°C
Time Frame: Measured during first 30 days from first dose of IMP.
Population: Participants with fever data reported
Measure: Mean (Standard Deviation); unit: Days
Units Other Than Participants: Days a temperature should be reported
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 293 | 293
Number analyzed (Days a temperature should be reported) | 4534 | 4558
Days | 20 (21.5) | 17.7 (20.2)

ADVERSE EVENTS:
Time Frame: Mortality and Symptomatic thrombotic events were assessed up to day 120; SAEs up to day 60
Arm/Group | Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 23/300 | 14/297
Serious Adverse Events (participants affected / at risk) | 77/300 | 82/297
Other Adverse Events (participants affected / at risk) | 8/300 | 5/297
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Arm (N=300) | Control Arm (N=297)
Sepsis (at least one event) (Infections and infestations) | 25 | 27
Organ Failure (at least one event) (General disorders) | 4 | 6
GvHD (at least one event) (Immune system disorders) | 5 | 7
Transfusion reaction (at least one event) (Blood and lymphatic system disorders) | 1 | 4
Fever (at least one event) (Infections and infestations) | 20 | 20
Other SAEs (at least one event) (General disorders) | 29 | 35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Arm (N=300) | Control Arm (N=297)
Venous thromboembolisms (Vascular disorders) | 7 | 4
Arterial ischaemic events (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/45/NCT03136445/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-13): https://cdn.clinicaltrials.gov/large-docs/45/NCT03136445/SAP_001.pdf